CLINICAL TRIAL: NCT05853835
Title: A Phase I First in Human, Randomized, Double-blind, Placebo- Controlled Study in Healthy Adult Volunteers to Evaluate Safety, Tolerability and Pharmacokinetics of LPX-TI641 After Single and Multiple Oral Doses.
Brief Title: First-in-Human Trial in Healthy Adult Volunteers to Evaluate Safety, Tolerability and PK of LAPIX Study Drug; LPX-TI641
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LAPIX Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LPX641-101
Record Dates: First submitted 2023-04-28; First posted 2023-05-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-06

CONDITIONS: Autoimmune Diseases; Multiple Sclerosis
MeSH Terms: conditions — Autoimmune Diseases; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigational drug blind will be maintained through a randomization schedule held by the dispensing pharmacist. The investigational drug blind shall not be broken by the site Investigator unless information concerning the investigational drug is necessary for the medical treatment of the subject. All study assessments and causality will be performed, if possible, prior to unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort-1 (Experimental): First dose of SAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort-2 (Experimental): Second dose of SAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort-3 (Experimental): Third dose of SAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort-4 (Experimental): Fourth dose of SAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort-5 (Experimental): Fifth dose of SAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort-6 (Experimental): Sixth dose of SAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort-7 (Experimental): First dose of MAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort 8 (Experimental): Second dose of MAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641
- Cohort 9 (Experimental): Third dose of MAD cohort (6 treatment + 2 placebo)
  Interventions: Drug: LPX-TI641

INTERVENTIONS:
Drug: LPX-TI641 — LAPIX Therapeutics Inc (LAPIX) has developed LPX-TI641, a small molecule for immune tolerance restoration/induction that is an orally bioavailable Tim family agonist (Tim-3 and Tim-4).

SUMMARY:
A Phase I First-in-Human, Randomized, Double-Blind, Placebo-Controlled Study in Healthy Adult Volunteers to Evaluate Safety, Tolerability, and Pharmacokinetics after Single and Multiple Oral Dose of LPX-TI641.

DETAILED DESCRIPTION:
This is a first-in-human, multi center, randomized, double-blinded, single and multiple ascending doses (SAD and MAD) Phase I study in healthy adult volunteers (HV).

The SAD cohorts will consist of six cohorts of eight participants (6 randomized to treatment + 2 randomized to placebo) in each cohort (Total 48 HV). Additional cohorts may be added.

The MAD cohorts will consist of 3 cohorts of eight participants (6 randomized to treatment + 2 randomized to placebo) in each cohort (Total 24 HV). The subjects in MAD cohorts will be dosed once daily for 7 consecutive days. Additional cohorts may be added.

Each entire cohort of 8 HV subjects will be enrolled at the same site.

ELIGIBILITY:
Inclusion Criteria: Healthy volunteers

1. Subject has signed an Informed Consent Form (ICF) prior to any study-specific procedures being performed
2. Healthy volunteers (HV) with no known acute or chronic medical conditions (respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, endocrine, etc.) at the time of enrollment.
3. Healthy volunteers (HV) with dermatological conditions are allowed if they are not receiving systemic treatments for their dermatological condition.
4. All male and non-pregnant females aged 18-55 years old irrespective of their race and ethnicity.
5. Body Mass Index (BMI) 18.0-30.0 kg/m2, inclusive at screening.
6. Clinical laboratory evaluations performed at screening, are within acceptable normal reference ranges (Grade 1 abnormalities may be acceptable if deemed necessary by the investigator. Grade 2 or higher would be exclusionary).
7. Subjects who are willing and able to adhere to study protocol requirements including but not limited to scheduled outpatient visits, inpatient hospital stay, laboratory tests, and 12-lead ECG.
8. Contraception - All subjects (male and female) must agree to use any two of the highly effective contraception methods listed below. This criterion must be followed from the time of the first dose of study medication for 6 weeks after the last dose in females and for 90 days after the last dose for males.

   a. The following applies to all female volunteers with childbearing potential and female partners of male volunteers enrolled in the study.

   i. Implantable progestogen-only hormone contraception associated with inhibition of ovulation.

ii. Intrauterine device. iii. Intrauterine hormone-releasing system. iv. Bilateral tubal occlusion. v. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: 1) Oral 2) Intravaginal 3)Transdermal 4) Injectable vi. Progestogen-only hormone contraception (oral or injectable) is associated with inhibition of ovulation.

vii. Vasectomized partner viii. Sexual abstinence -this is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated about the duration of the study and the preferred and usual lifestyle of the participant.

b. The following applies to all male subjects in the study: i. Sexual abstinence- this is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated for the duration of the study and the preferred and usual lifestyle of the participant.

ii. A combination of male condoms with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods).

iii. Vasectomy

Exclusion Criteria: Healthy volunteers

1. Any known history of malignancy
2. Any known history of asthma
3. COVID-19:

   The subject has COVID-19 positive status (confirmed by clinical signs and symptoms and a positive SARS-CoV-2 NAAT result COVID test) at any time during the screening period.

   OR has had recent COVID-19 vaccination including a booster dose in the past 30 days

   OR has received anti-viral therapy intended to prevent COVID-19 such as nelmetavir/ritonavir, remdesivir, molnupiravir, interferons, Anti-SARS-CoV-2 monoclonal antibodies, IVIG SARS-CoV-2, COVID-19 Convalescent plasma, etc. within the past 30 days
4. Subject with positive results for HBsAg (hepatitis B surface antigens) and/or HBcAb (Hepatitis B core antibodies) and/or HCV Ab (hepatitis C antibodies), and/or HIV Ab (human immunodeficiency virus antibodies).
5. Blood loss of >250 mL or donated blood within 56 days or donated plasma within 7 days of screening.
6. Recent vaccination with live attenuated vaccines such as influenza, MMR, Herpes zoster, varicella, yellow fever, Rotavirus vaccine, etc., or inactivated vaccines such as Hepatitis A, Rabies vaccine, etc. in the past 30 days.
7. Abnormal amylase levels (Grade 2 or greater)
8. Clinically significant ECG abnormalities (QTcF >450 ms for males and QTcF >470 ms for females).
9. History of or current compulsive abuse of alcohol or positive test for alcohol at screening or Day 0 of Visit 1
10. History of or current use of or positive test at screening or Day 0 of Visit 1 for drugs such as marijuana, cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives.
11. Consumption of any beverages or food containing alcohol or drugs such as marijuana, cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives from screening until donating the last sample of the study
12. Use of medications for the timeframes specified below, except for medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    * prescription medications within 14 days prior to dosing or 5 half-lives, whichever is longer;
    * over-the-counter products and natural health products (including herbal remedies homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 14 days prior to dosing or 5 half-lives, whichever is longer, except for the occasional use of paracetamol (up to 2 g daily);
    * any prescription or over-the-counter medication or natural health products used for the treatment of irregular bowel transit (e.g,. diarrhea, constipation) within 4 weeks prior to dosing;
    * depot injection or implant of any drug within 3 months prior to dosing;
    * use of any drugs known to induce or inhibit hepatic metabolism (including St. John's Wort [hypericin]) within 14 days prior to dosing.
13. The subject has participated in another investigational study involving any investigational product within 60 days, or 5 half-lives, whichever is longer, before the dose of the study drug.
14. Pregnant or lactating women or women currently undergoing infertility treatments or women who intend to become pregnant during the time of study enrollment.
15. Involvement in the planning and conduct of the study (applies to CRO staff or staff at the study site).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability after single ascending oral doses of LPX-TI641 in healthy adult volunteers. | 14 days
  Proportion of subjects with AEs, SAEs and DLTs will be recorded.
To evaluate the safety and tolerability after multiple ascending oral doses of LPX-TI641 in healthy adult volunteers. | 21 days
  Proportion of subjects with AEs, SAEs and DLTs will be recorded.

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics after single ascending oral doses of LPX-TI641 in healthy adult volunteers. | Day 1
  Measurements of PK parameters including
  * Maximum observed plasma concentration (Cmax),
  * Time to first occurrence of Cmax (Tmax),
  * Area under the plasma concentration-time curve from time 0 to the time last concentration measurement (AUC0-last)
  * Area under the plasma concentration-time curve from time 0 to 24 hr (AUC0-24)
  * Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞),
  * Percentage AUC extrapolated (%AUCextrap)
  * Terminal disposition phase half-life (t1/2z),
  * Apparent clearance after extravascular administration (CL/F),
  * Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F)
To evaluate the plasma pharmacokinetics after multiple ascending oral doses of LPXTI641 in healthy adult volunteers. | Day 1 and Day 7
  Measuring the PK parameters such as Cmax, Tmax, AUC0-last, AUC0-24, %AUCextrap, t1/2, CL/F, Vz/F at steady state
  * Minimal observed concentration within the dosing interval (Ctrough)
  * Accumulation index (Cmax and AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Mahmoud Shennak, MD, Principal Investigator — Triumpharma; John Mickelson, DO, Principal Investigator — AXIS Clinicals, Dilworth, Minnesota USA
Locations (2):
- AXIS Clinicals, Dilworth, Minnesota, United States
- Triumpharma clinical research unit at Alessra Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No